CLINICAL TRIAL: NCT01083173
Title: Post-Marketing Surveillance of Safety and Efficacy of Kaletra® Tablet in Korean Patients Under the "New Drug Re-Examination"
Brief Title: Surveillance of Kaletra in Korean Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P11-068
Record Dates: First submitted 2010-02-19; First posted 2010-03-09 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
Keywords: Postmarketing Drug Surveillance; HIV-1 infection; Kaletra

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with HIV-1 infection: Participants treated with Kaletra (lopinavir/ritonavir 200 mg/50 mg and 100 mg/25 mg) tablet

SUMMARY:
This single-arm, multi-center, Post-Marketing Surveillance study of Kaletra (lopinavir/ritonavir) was conducted in accordance with the approved Korean product labeling in participants 2 years of age and older with human immunodeficiency virus type 1 (HIV-1) infection.

DETAILED DESCRIPTION:
Participants were observed for up to 48 weeks following the first dose of Kaletra. A follow-up visit took place 1-2 weeks after treatment initiation, and subsequent visits occurred at the discretion of the investigators, typically occurring every 3 months. Clinical/immunological/virological/laboratory status, Kaletra-containing regimen/concomitant medication information, and adverse event information were obtained at follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients 2 years of age and above with HIV-1 infection
* Patients who were prescribed Kaletra treatment as per investigator's medical judgment
* Patients who gave verbal or written authorization to use their personal and health data
* Patients who started Kaletra treatment after study agreement was in place

Exclusion Criteria:

* Patients with known hypersensitivity to lopinavir, ritonavir or any excipients of the Kaletra tablet
* Patients who were being treated or will be treated with drugs that are contraindicated with Kaletra
* Patients who have been treated with Kaletra
* Patients participating in other clinical trials

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: general hospitals
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2009-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SoRa Lee, MD, Study Director — AbbVie Ltd.

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Surveillance: The safety population included all participants who received at least one dose of Kaletra, and the effectiveness population included all participants who received Kaletra treatment for at least 24 weeks.
- Long-term Surveillance: The safety population included all participants who received Kaletra for more than 24 weeks, and the effectiveness population included all participants who received Kaletra treatment for at least 48 weeks.
Period: Main Surveillance: Safety Group
Arm/Group | Main Surveillance | Long-term Surveillance
Started | 595 | 0
Completed | 580 | 0
Not Completed | 15 | 0
Not completed — Violation of inclusion/exclusion crit. | 14 | 0
Not completed — Violation of the use/dosage | 1 | 0
Period: Main Surveillance: Effectiveness Group
Arm/Group | Main Surveillance | Long-term Surveillance
Started | 580 | 0
Completed | 198 | 0
Not Completed | 382 | 0
Not completed — No follow-up at 24 ±4 wks | 201 | 0
Not completed — No viral load data at 24 ±4 wks | 168 | 0
Not completed — Administration of Kaletra <24 wks | 13 | 0
Period: Long-term Surveillance: Safety Group
Arm/Group | Main Surveillance | Long-term Surveillance
Started | 0 | 595
Completed | 0 | 479
Not Completed | 0 | 116
Not completed — Violation of inclusion/exclusion crit. | 0 | 14
Not completed — Violation of the dosage | 0 | 1
Not completed — Administration of Kaletra <20 wks | 0 | 101
Period: Long-term Surveillance: Effectiveness Gr
Arm/Group | Main Surveillance | Long-term Surveillance
Started | 0 | 479
Completed | 0 | 102
Not Completed | 0 | 377
Not completed — No follow-up at 48 ±4 wks | 0 | 195
Not completed — No viral load data at 48 ±4 wks | 0 | 136
Not completed — Administration of Kaletra <48 wks | 0 | 46

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: The main surveillance safety population included all participants who received at least one dose of Kaletra. The long-term surveillance safety population included participants who received Kaletra for more than 24 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 580
Age, Customized [Mean (Standard Deviation); unit: years]
  Main Surveillance n= 580 | 41.3 (12.5)
  Long-term Surveillance n=479 | 41 (12.1)
Sex/Gender, Customized [Number; unit: participants]
  Main Surveillance Females | 56
  Main Surveillance Males | 524
  Long-Term Surveillance Females | 47
  Long-Term Surveillance Males | 432

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events were recorded during the 48-week surveillance period and until 30 days following the last dose.
Time Frame: From the start of treatment until 30 days after the last dose, up to 52 weeks
Population: Participants with available data
Measure: Number; unit: participants
Groups:
- Main Surveillance: All participants who received at least one dose of Kaletra
- Long-term Surveillance: Participants who received Kaletra for more than 24 weeks
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 580 | 479
participants | 363 | 285

2. Primary Outcome: Number of Participants Who Interrupted or Discontinued Kaletra Treatment
Description: At 24 and 48 weeks after initiation of Kaletra treatment or upon permanent discontinuation of Kaletra treatment, the investigator documented Kaletra status (on-going, permanently discontinued, lost to follow-up, etc).
Time Frame: Weeks 24 and 48 after initiation of Kaletra treatment or upon permanent discontinuation of Kaletra treatment
Population: Participants with available data
Measure: Number; unit: participants
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 580 | 479
participants | 120 | 43

3. Primary Outcome: Percentage of Participants With Viral Load Below 400 Copies/mL
Description: Blood samples were obtained from participants 24 weeks after the start of Kaletra treatment, and analyzed for human immunodeficiency virus-1 (HIV-1) RNA levels.
Time Frame: Week 24
Population: Participants with available data
Measure: Number; unit: percentage of participants
Groups:
- Main Surveillance: All participants who received Kaletra treatment for at least 24 weeks
Arm/Group | Main Surveillance
Number analyzed (Participants) | 198
percentage of participants | 92.4

4. Secondary Outcome: Change From Baseline in Viral Load
Description: This variable, change from baseline in viral load, was not included in the final protocol. Therefore, these data were not calculated.
Time Frame: Week 24 & 48
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Counts
Description: Blood samples were obtained from participants at baseline, 24, and 48 weeks after the start of Kaletra treatment and analyzed for CD4 cell counts. Change in CD4 cell counts in the main surveillance population was calculated by subtracting the value at baseline from the value at 24 weeks. Change in CD4 cell counts in the long-term surveillance population was calculated by subtracting the value at baseline from the value at 48 weeks.
Time Frame: From baseline to Weeks 24 and 48
Population: Participants with available data
Measure: Mean (Standard Deviation); unit: cells/mm˄3
Groups:
- Long-term Surveillance: All participants who received Kaletra treatment for at least 48 weeks
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 181 | 93
cells/mm˄3 | 145.47 (144.28) | 170.47 (159.30)
Statistical Analysis 1: Comparison: Main Surveillance; CD4 cell counts at 24 weeks as compared to baseline; Test type: Superiority or Other; p < 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Long-term Surveillance; CD4 cell counts at 48 weeks as compared to baseline; Test type: Superiority or Other; p < 0.0001, Paired t-test

6. Secondary Outcome: Percentage of Participants With Confirmed Viral Resistance
Description: Blood samples were obtained from participants at initiation of Kaletra treatment and follow up visits through weeks 24 and 48 and analyzed for genotypic viral resistance.
Time Frame: From baseline through weeks 24 and 48
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 198 | 102
percentage of participants | 0.51 | 1.96

7. Secondary Outcome: Mean Time to Treatment Failure
Description: Blood samples were obtained from participants at initiation of Kaletra treatment and at follow up visits through weeks 24 and 48 and analyzed for human immunodeficiency virus-1 (HIV-1) RNA levels. Treatment failure was defined as HIV RNA level > 400 copies/mL at week 24 and HIV RNA level > 50 copies/mL at week 48.
Time Frame: From baseline through weeks 24 and 48
Population: Participants with available data
Measure: Mean (Standard Error); unit: days
Arm/Group | Main Surveillance | Long-term Surveillance
Number analyzed (Participants) | 198 | 102
days | 399.97 (3.45) | 410.8 (1.03)

8. Primary Outcome: Percentage of Participants With Viral Load Below 50 Copies/mL
Description: Blood samples were obtained from participants 48 weeks after the start of Kaletra treatment, and analyzed for human immunodeficiency virus-1 (HIV-1) RNA levels.
Time Frame: Week 48
Population: Participants with available data
Measure: Number; unit: percentage of participants
Arm/Group | Long-term Surveillance
Number analyzed (Participants) | 102
percentage of participants | 68.6

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the last dose, up to 52 weeks
Description: Adverse event(s) details, including the type of adverse event(s), onset/end date, severity, action taken, and relationship to the drug and the investigator's view on the adverse event(s) (whether it was related to the drug or not) were recorded during the 48-week surveillance period and until 30 days following the last dose.
Arm/Group | Main Surveillance | Long-term Surveillance
Serious Adverse Events (participants affected / at risk) | 51/580 | 39/479
Other Adverse Events (participants affected / at risk) | 222/580 | 169/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Main Surveillance (N=580) | Long-term Surveillance (N=479)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 3 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Retinal detachment (Eye disorders) | 1 | 1
Retinal haemorrhage (Eye disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 2
Chest discomfort (General disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1
Herpes zoster (Infections and infestations) | 5 | 5
Pneumocystis jirovecii pneumonia (Infections and infestations) | 8 | 5
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 4 | 3
Progressive multifocal leukoencephalopathy (Infections and infestations) | 2 | 1
Disseminated tuberculosis (Infections and infestations) | 1 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 2
Arthritis bacterial (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Mycobacterial infection (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 1
Spleen tuberculosis (Infections and infestations) | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Depression (Psychiatric disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Main Surveillance (N=580) | Long-term Surveillance (N=479)
Diarrhoea (Gastrointestinal disorders) | 119 | 88
Nausea (Gastrointestinal disorders) | 70 | 49
Nasopharyngitis (Infections and infestations) | 33 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.